CLINICAL TRIAL: NCT06590220
Title: Establishment of Multiparametric Prediction Models for Moderate to Severe Thyroid Associated Ophthalmopathy
Brief Title: Establishment of Multiparametric Prediction Models for Moderate to SevereThyroid Associated Ophthalmopathy
Status: Recruiting | Type: Observational
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Tuo Li, MD, Deputy Director, Shanghai Changzheng Hospital
Other Study IDs: TAO3M-2
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Thyroid Associated Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TAO

SUMMARY:
Thyroid-associated ophthalmopathy (TAO) is an organ-specific autoimmune disease closely related to thyroid disease, which leads the incidence of orbital disease in adults and is the most common cause of diffuse toxic goiter (Graves disease, GD). The clinical manifestations of TAO are complex and varied. In severe cases, it may seriously impair visual function, affect daily life, and even cause corneal ulceration, perforation, and blindness. Therefore, a reasonable and effective treatment plan should be chosen according to the degree of TAO.

The aim of this clinical study is to:

1. Found the new diagnostic markers or imaging sequences.
2. Establish and validate a multimodal and multiparameter prediction model for moderate to severe TAO.

ELIGIBILITY:
Inclusion Criteria:

* According to the Bartley criteria，diagnosed TAO at our hospital after 2024/8/31
* Moderate to severe patients defined by EUGOGO
* CAS ≥3 (on the 7-item scale) for the study eye

Exclusion Criteria:

* Anticipated need for intervention due to sight-threatening complications or other significant and acute deterioration in vision
* History of systemic (eg, oral or IV) steroid use with a cumulative dose equivalent to >1 g of methylprednisolone for the treatment of TAO.
* Any major illness/condition or evidence of an unstable clinical condition that, in the investigator's judgment, will substantially increase the risk to the participant, or confound the interpretation of safety assessments, if they were to participate in the study
* Any other condition that, in the opinion of the investigator, would impair the ability of the participant to comply with the study procedures or impair the ability to interpret data from the participant's participation in the study
* Pregnant or lactating
* Any other condition that,would impair the ability of the participant to undergo orbital MRI
* Incomplete information

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Moderate to severe active TAO patients who receive medical treatment and assessment
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-09-06 (Estimated); Study Completion 2028-09-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with overall response | 1 week after the end of treatment
Percentage of participants with overall response | 24 weeks after the end of treatment
Percentage of participants with overall response | 52 weeks after the end of treatment
Percentage of participants with overall response | 104 weeks after the end of treatment

SECONDARY OUTCOMES:
Incidence and characterization of nonserious treatment emergent adverse events (TEAEs) | 1 week after the end of treatment
  Safety and Tolerability
Change of Serum Lipids parameters from baseline | 104 weeks after the end of treatment
  including TG（mmol/L）、TC（mmol/L）、HDL（mmol/L）、LDL（mmol/L）
Change of Serum T3、T4 level from baseline | 104 weeks after the end of treatment
  including T3（nmol/L）、T4（nmol/L）
Change of Serum TSH level from baseline | 104 weeks after the end of treatment
  including TSH（mIU/L）
Change of Serum FT3、FT4 level from baseline | 104 weeks after the end of treatment
  including FT3（pmol/L）、FT4（pmol/L）
Change of Serum TRAb from baseline | 104 weeks after the end of treatment
  including TRAb（IU/l）

OTHER OUTCOMES:
change of extraocular muscle volume and orbital fat volume by MRI | 104 weeks after the end of treatment
Change of Serum T-cell subgroup | 1 week after the end of treatment
  including CD3（%）、CD3 absolute value、CD4（%）、CD4 absolute value、CD8（%）、CD8 absolute value、CD4/CD8（%）
Change of Serum T-cell subgroup | 104 weeks after the end of treatment
  including CD3（%）、CD3 absolute value、CD4（%）、CD4 absolute value、CD8（%）、CD8 absolute value、CD4/CD8（%）
change of extraocular muscle volume and orbital fat volume by MRI | 4 weeks after the end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhai L, Luo B, Wu H, Wang Q, Yuan G, Liu P, Ma Y, Zhao Y, Zhang J. Prediction of treatment response to intravenous glucocorticoid in patients with thyroid-associated ophthalmopathy using T2 mapping and T2 IDEAL. Eur J Radiol. 2021 Sep;142:109839. doi: 10.1016/j.ejrad.2021.109839. Epub 2021 Jul 3. PMID 34252869
- [Background] Cevik Y, Taylan Sekeroglu H, Ozgen B, Erkan Turan K, Sanac AS. Clinical and Radiological Findings in Patients with Newly Diagnosed Graves' Ophthalmopathy. Int J Endocrinol. 2021 Apr 30;2021:5513008. doi: 10.1155/2021/5513008. eCollection 2021. PMID 34007271